CLINICAL TRIAL: NCT04650802
Title: Improving Propulsion of the Paretic Leg In Chronic Stroke
Acronym: I-PICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 785_LOPES I-PICS; R201605453 (Other Grant/Funding Number: Revalidatiefonds)
Record Dates: First submitted 2020-11-13; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Stroke
Keywords: Gait; Rehabilitation; Robotics; Propulsion; Speed; Biomechanics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Longitudinal intervention study with two consecutive baseline assessments and a five-week follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gait training (Experimental): Participants receive five weeks individual robotic gait training in LOPES II, targeting paretic propulsion (60 minutes, two time a week). The robotic gait training is complemented with daily home exercises (15 minutes/day) focusing on increasing strength and practice of learned strategies in daily life.
  Interventions: Device: Gait training

INTERVENTIONS:
Device: Gait training — Participants receive five weeks individual robotic gait training in LOPES II, targeting paretic propulsion (60 minutes, two time a week). The robotic gait training is complemented with daily home exercises (15 minutes/day) focusing on increasing strength and practice of learned strategies in daily life.

SUMMARY:
Stroke survivors may have a latent, propulsive capacity of the paretic leg, that can be elicited during short, intensive gait training interventions. The aim of this study was therefor to investigate the effect of a five-week gait training on paretic propulsion, propulsion symmetry, gait capacity, and daily-life mobility and physical activity in chronic stroke survivors.

DETAILED DESCRIPTION:
Stroke survivors may have a latent, propulsive capacity of the paretic leg, that can be elicited during short, intensive gait training interventions. The aim of this study was therefor to investigate the effect of a five-week gait training on paretic propulsion, propulsion symmetry, gait capacity, and daily-life mobility and physical activity in chronic stroke survivors. We hypothesize that the robotic gait training will improve propulsion symmetry and, thereby, gait speed and functional gait tasks. In addition, we expect that improved gait capacity might lead to less impact of stroke on daily-life mobility and a higher physical activity level. Thirty-three chronic stroke survivors with impaired paretic propulsion (≥8% difference in paretic vs. non-paretic propulsive impulse) will be enrolled in this proof-of-concept study. Participants receive five weeks individual robotic gait training targeting paretic propulsion (60 minutes, two time a week). The robotic gait training is complemented with daily home exercises (15 minutes/day) focusing on increasing strength and practice of learned strategies in daily life. Propulsion measures, self-selected gait speed, performance on functional gait tasks, and daily-life mobility and physical activity are assessed five weeks (T0) and one week (T1) before the start of the intervention, and one week (T2) and five weeks (T3) after the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* adults (>18 years of age) with unilateral ischemic or heamorrhagic supratentorial stroke
* at least 6 months post-onset
* impaired propulsion of the paretic leg during walking at a self-selected speed (≥ 8 percent propulsion asymmetry)
* ability to walk 10 meter without support or use of a walking aid (Functional Ambulatory Categories (FAC) 3-5)
* ability to walk for 5 consecutive minutes, with or without the use of a walking aid
* at least 10 degrees passive hip extension and able to stand plantigrade with extended knee

Exclusion Criteria:

* inability to move the body upward against gravity (calf muscle - Medical Research Council (MRC) scale < 3)
* severe cognitive problems assessed with Mini-Mental State Examination (MMSE < 24)
* depressed mood assessed with the Hospital Anxiety and Depression Score (HADS > 7)
* persistent unilateral visuospatial neglect assessed with the Star Cancellation Test (score < 44)
* any medical condition interfering with gait
* inability to understand verbal instructions
* inappropriate or unsafe fitting of the robotic gait trainer, due to severe lower limb spasticity (Modified Ashworth Scale (MAS) ≥ 3), severe lower limb contractures, body weight ≥ 140 kg, or skin problems at body sites where the harness or straps were to be fitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Change in propulsion symmetry at self-selected gait speed between pre- and post-intervention | Assessments are performed five weeks (T0) and one week (T1) before the start of the intervention, and one week (T2) and five weeks (T3) after the end of the five-week intervention period.
  Propulsion symmetry was calculated by dividing the paretic propulsive impulse by the sum of the paretic and non-paretic propulsive impulse

SECONDARY OUTCOMES:
Change in self-selected gait speed between pre- and post-intervention | Assessments are performed five weeks (T0) and one week (T1) before the start of the intervention, and one week (T2) and five weeks (T3) after the end of the five-week intervention period.
  Participants walked at their self-selected, comfortable speed along a straight six-meter walkway. Gait speed was determined in m/s.
Change in trailing limb angle of the paretic leg between pre- and post-intervention | Assessments are performed five weeks (T0) and one week (T1) before the start of the intervention, and one week (T2) and five weeks (T3) after the end of the five-week intervention period.
  The position of the hip joint center and toe marker, determined with a 3D gait analysis, were used to calculate the trailing limb angle (in degrees) of the paretic leg at the instant of peak paretic anterior ground reaction force.
Change in ankle plantarflexion moment of the paretic leg between pre- and post-intervention | Assessments are performed five weeks (T0) and one week (T1) before the start of the intervention, and one week (T2) and five weeks (T3) after the end of the five-week intervention period.
  Vicon Plug-In-Gait model and software were used to calculate paretic ankle plantarflexion moment (Nm/kg) at the instant of peak paretic anterior ground reaction force.
Change in performance on the Six-minute walk test between pre- and post-intervention | Assessments are performed five weeks (T0) and one week (T1) before the start of the intervention, and one week (T2) and five weeks (T3) after the end of the five-week intervention period.
  Six-minute walk test (meters) was performed.
Change in performance on the Functional gait assessment between pre- and post-intervention | Assessments are performed five weeks (T0) and one week (T1) before the start of the intervention, and one week (T2) and five weeks (T3) after the end of the five-week intervention period.
  Functional gait assessment (score range 0-30) was performed. Higher scores indicate better outcome.
Change in daily-life mobility between pre- and post-intervention | Assessments are performed five weeks (T0) and one week (T1) before the start of the intervention, and one week (T2) and five weeks (T3) after the end of the five-week intervention period.
  Daily-life mobility was assessed with the Stroke Impact Scale (SIS - domain Mobility, range 0-100). Higher scores indicate better outcome.
Change in daily-life physical activity between pre- and post-intervention | Assessments are performed five weeks (T0) and one week (T1) before the start of the intervention, and one week (T2) and five weeks (T3) after the end of the five-week intervention period.
  Daily-life physical activity was assesed using an activity-tracker (Activ8). Participants wore the activity tracker for 24 hours a day, for a minimum of five consecutive days. Total time of walking and the intensity of walking were determined.
Static postural balance at baseline | Assessments are performed five weeks (T0) before the start of the intervention.
  To determine the association between individuals' baseline characteristics and the training response the determinant was assessed during stance using forceplates at T0.
The difference in propulsion impulse of the paretic leg during walking at fast vs. self-selected speed at baseline | Assessments are performed five weeks (T0) before the start of the intervention.
  To determine the association between individuals' baseline characteristics and the training response the determinant was assessed during the 3D-gait analysis at T0.
Maximal ankle plantarflexion moment at baseline | Assessments are performed five weeks (T0) before the start of the intervention.
  To determine the association between individuals' baseline characteristics and the training response the determinant was assessed with the Biodex at T0.
Score on the maximal steplength test at baseline | Assessments are performed five weeks (T0) before the start of the intervention.
  To determine the association between individuals' baseline characteristics and the training response the determinant was assessed at T0.

CONTACTS AND LOCATIONS:
Overall Officials: ACH Geurts, Prof. dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Sint Maartenskliniek, Ubbergen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alingh JF, Groen BE, Kamphuis JF, Geurts ACH, Weerdesteyn V. Task-specific training for improving propulsion symmetry and gait speed in people in the chronic phase after stroke: a proof-of-concept study. J Neuroeng Rehabil. 2021 Apr 23;18(1):69. doi: 10.1186/s12984-021-00858-8. PMID 33892754